CLINICAL TRIAL: NCT00336856
Title: A Phase 2 Study of Irinotecan and Cetuximab on an Every 2 Week Schedule, as Second Line Therapy in Patients With Advanced Colorectal Cancer
Brief Title: Irinotecan and Cetuximab for Colorectal Cancer as Second Line Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Nathan Bahary, MD, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-006
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Colon Cancer; Rectum Cancer
Keywords: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IRINOTECAN AND CETUXIMAB (Experimental): Cetuximab will be administered at the dose of 500 mg/m2 intravenously (IV) over 120 minutes, followed by 500 mg/m2 every 2 weeks, IV over 2 hours at an infusion rate not to exceed 5 ml/min. Followed immediately by Irinotecan administered at a dose of 180 mg/m2 IV over 60 minutes every two weeks.
  Interventions: Drug: Cetuximab; Drug: Irinotecan

INTERVENTIONS:
Drug: Cetuximab — The treatment will include cetuximab 500 mg/m² IV for 120 minutes followed by irinotecan 180 mg/m² or 60 minutes. The starting dose of irinotecan for patients who are 70 years old or greater, or who have had radiation therapy to the abdomen or pelvis, or whose level of functioning is poor (performance status of 2) will have a starting dose of 150 mg/m2 for irinotecan. All subsequent treatments will include cetuximab 500 mg/m² IV over 60 minutes and irinotecan 150 mg/m² or 180 mg/m2 intravenously over 60 minutes every 2 weeks.
Drug: Irinotecan — The treatment will include cetuximab 500 mg/m² IV for 120 minutes followed by irinotecan 180 mg/m² or 60 minutes. The starting dose of irinotecan for patients who are 70 years old or greater, or who have had radiation therapy to the abdomen or pelvis, or whose level of functioning is poor (performance status of 2) will have a starting dose of 150 mg/m2 for irinotecan. All subsequent treatments will include cetuximab 500 mg/m² IV over 60 minutes and irinotecan 150 mg/m² or 180 mg/m2 intravenously over 60 minutes every 2 weeks.

SUMMARY:
Research Hypothesis: Subjects in the study population who are treated with cetuximab in combination with irinotecan will have higher response rates than subjects treated with irinotecan alone.

DETAILED DESCRIPTION:
Primary Objective:

·The primary aim of this study is to assess the response rate of patients with previously treated colorectal cancer (CRC) Number of Subjects: 31

Study Population:

Subjects with metastatic, CRC who have failed a first-line chemotherapeutic regimen containing oxaliplatin and a fluoropyrimidine, and who have not previously received irinotecan or cetuximab for treatment of CRC.

Test Product, Dose and Mode of Administration, Duration of Treatment:

Cetuximab administered at an initial dose of 500 mg/m2 intravenously (IV) over 120 minutes, followed by 500 mg/m2 every 2 weeks IV over 60 minutes.

Reference Therapy, Dose and Mode of Administration, Duration of Treatment: Irinotecan administered at a dose of 150a or 180 mg/m2 IV over 60 minutes every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must consent to be in the study
* Patients must have advanced, surgically unresectable CRC, who have failed a first line metastatic regimen, within 12 months of starting protocol therapy.
* Patients must have measurable disease
* There must be histologic confirmation of adenocarcinoma of the colon or rectum.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Estimated life expectancy of at least 12 weeks.
* One prior therapy for metastatic disease is permitted.
* Recurrence within 12 months of adjuvant therapy with FOLFOX or a similar regimen (i.e FLOX, CapOX) is considered one regimen and allowed for study
* There must be evidence of adequate organ function
* Patients with a history of prior non-colorectal malignancies are eligible if they have been disease-free for ³ 5 years prior to study entry and are deemed by the physician to be at low risk for recurrence.
* Age > 18 yrs.

Exclusion Criteria:

* Any prior therapy with irinotecan or cetuximab or an EGFR targeting agent.
* Any systemic therapy administered for metastatic or locally recurrent colorectal cancer within 28 days of study treatment.
* Patients who are considered candidates for surgical resection of metastatic and/or locally advanced disease.
* Any histology other than adenocarcinoma of the colon or rectum.
* Serious concomitant medical conditions that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study.
* Evidence of central nervous system metastases
* Pulmonary fibrosis or interstitial pneumonitis
* General Medical Concerns
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
* Serious, uncontrolled, concurrent infection.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study; fine needle aspirations or core biopsies within 7 days prior to Day 0. Line placement (i.e Infus-a-port or PICC) is not considered major surgery.
* Evidence of bleeding diathesis or coagulopathy
* Prior severe infusion reaction to a monoclonal antibody.
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* Patients with Gilbert's Syndrome
* Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.
* All WOCBP MUST have a negative pregnancy test within 7 days prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study.
* In addition, all WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
* The Investigator must immediately notify BMS in the event of a confirmed pregnancy in a patient participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Bahary, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Centers, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- IRINOTECAN AND CETUXIMAB: Subjects with metastatic, CRC who have failed a first-line chemotherapeutic regimen containing oxaliplatin and a fluoropyrimidine, and who have not previously received irinotecan or cetuximab for treatment of CRC
Period: Overall Study
Arm/Group | IRINOTECAN AND CETUXIMAB
Started | 35 (Number of patients consented and registered for the study)
Completed | 31
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Found ineligible at time of analysis | 1

BASELINE CHARACTERISTICS:
Population: Patients who received at least one dose of Irinotecan administered at a dose of 150a or 180 mg/m2 IV every two weeks, were thus evaluable and included in outcome analyses.
Groups:
- IRINOTECAN AND CETUXIMAB: Subjects with metastatic, CRC who have failed a first-line chemotherapeutic regimen containing oxaliplatin and a fluoropyrimidine, and who have not previously received irinotecan or cetuximab for treatment of CRC who received Cetuximab administered at an initial dose of 500 mg/m2 intravenously (IV), followed by 500 mg/m2 every 2 weeks IV
Arm/Group | IRINOTECAN AND CETUXIMAB
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 61.8 [43 to 83.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: Percentage of partial responses (PR) + complete responses (CR).
Time Frame: every 6 - 8 weeks, up to 30 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- IRINOTECAN AND CETUXIMAB: Cetuximab administered at an initial dose of 500 mg/m2 intravenously (IV) over 120 minutes, followed by 500 mg/m2 every 2 weeks IV over 60 minutes.
  Irinotecan administered at a dose of 150 or 180 mg/m2 IV over 60 minutes every two weeks.
Arm/Group | IRINOTECAN AND CETUXIMAB
Number analyzed (Participants) | 31
percentage of participants | 6 [0.79 to 21]

2. Secondary Outcome: Time to Progression
Description: time from start of protocol therapy until objective tumor progression
Time Frame: Up to 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IRINOTECAN AND CETUXIMAB
Number analyzed (Participants) | 31
months | 2.4 [1.3 to 4.6]

3. Secondary Outcome: Overall Survival
Description: time from start of protocol therapy until death from any cause
Time Frame: Up to 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IRINOTECAN AND CETUXIMAB
Number analyzed (Participants) | 31
months | 9.3 [5.1 to 15]

ADVERSE EVENTS:
Arm/Group | IRINOTECAN AND CETUXIMAB
Serious Adverse Events (participants affected / at risk) | 13/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IRINOTECAN AND CETUXIMAB (N=32)
Lymphopenia (Investigations) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Supraventricular and nodal arrhythmia, Atrial fibrillation (Cardiac disorders) | 1
Cardiac General - Other (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1
Constitutional Symptoms - Other (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10^9 cells/L) (General disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fistula, GI, Abdomen NOS (Gastrointestinal disorders) | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Obstruction, GI, Colon (Gastrointestinal disorders) | 2
Perforation, GI, Ileum (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils, Abdomen NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Wound (Infections and infestations) | 1
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 1
Alkaline phosphatase (Metabolism and nutrition disorders) | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Pain, Abdomen NOS (Gastrointestinal disorders) | 3
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IRINOTECAN AND CETUXIMAB (N=32)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
Alkaline phosphatase (Metabolism and nutrition disorders) | 1
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 13
Ascites (non-malignant) (Gastrointestinal disorders) | 2
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 21
Distension/bloating, abdominal (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 3
Dry eye syndrome (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8
Edema: limb (General disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 22
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9 cells/L) (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 5
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 11
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 10
Hemorrhage, GI, Lower GI NOS (Gastrointestinal disorders) | 1
Hemorrhage, GI, Rectum (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection - Other (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Bladder (urinary) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Blood (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Skin (cellulitis) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Upper airway NOS (Infections and infestations) | 3
Infection with normal ANC or Grade 1 or 2 neutrophils, Urinary tract NOS (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils, Vulva (Infections and infestations) | 1
Injection site reaction/extravasation changes (General disorders) | 1
Insomnia (Psychiatric disorders) | 1
Leukocytes (total WBC) (Investigations) | 11
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1
Memory impairment (Nervous system disorders) | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1
Mood alteration, Anxiety (Psychiatric disorders) | 1
Mood alteration, Depression (Psychiatric disorders) | 1
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 8
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 13
Neurology - Other (Nervous system disorders) | 4
Neuropathy: motor (Nervous system disorders) | 4
Neuropathy: sensory (Nervous system disorders) | 9
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 9
Obstruction, GI, Small bowel NOS (Gastrointestinal disorders) | 2
Ocular/Visual - Other (Eye disorders) | 1
Pain - Other (General disorders) | 2
Pain, Abdomen NOS (Gastrointestinal disorders) | 10
Pain, Back (Musculoskeletal and connective tissue disorders) | 4
Pain, Chest/thorax NOS (General disorders) | 1
Pain, Extremity-limb (Musculoskeletal and connective tissue disorders) | 2
Pain, Middle ear (Ear and labyrinth disorders) | 1
Pain, Rectum (Gastrointestinal disorders) | 1
Platelets (Investigations) | 2
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 19
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4
Renal failure (Renal and urinary disorders) | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 2
Rigors/chills (General disorders) | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1
Supraventricular and nodal arrhythmia, Sinus bradycardia (Cardiac disorders) | 1
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3
Ulcer, GI, Stomach (Gastrointestinal disorders) | 1
Ulceration (General disorders) | 1
Vitreous hemorrhage (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight gain (Investigations) | 1
Weight loss (Investigations) | 5
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes